CLINICAL TRIAL: NCT02107586
Title: Biceps Tenotomy or Tenodesis in Treating Long Head of the Biceps Pathology: a Prospective Randomized Controlled Trial
Brief Title: Comparison of Outcomes Between Biceps Tenotomy and Tenodesis in the Treatment of the Long Head of the Biceps Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-0117
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Chronic Refractive Bicipital Pain
Keywords: biceps tenodesis; biceps tenotomy; biceps tendonitis; biceps inflammation; shoulder surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biceps tenodesis (Active Comparator): 32 subjects in the study will receive biceps tenodesis as a surgical intervention
  Interventions: Procedure: Biceps tenodesis
- Biceps tenotomy (Active Comparator): 32 subjects in the study will receive biceps tenotomy as a surgical intervention
  Interventions: Procedure: Biceps tenotomy

INTERVENTIONS:
Procedure: Biceps tenotomy — A biceps tenotomy procedure involves cutting of the long head of the biceps just prior to its insertion on the superior labrum of the glenoid.
  Arms: Biceps tenotomy
Procedure: Biceps tenodesis — Biceps tenodesis involves detaching the long head of the biceps from it's superior labrum in the shoulder and reattaching it to the humerus bone just below the shoulder.
  Arms: Biceps tenodesis

SUMMARY:
The purpose of the study is to determine what the different outcomes are for biceps tenodesis and tenotomy in the treatment of the long head of the biceps pathology.

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic refractive bicipital pain

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2014-04-08 (Actual); Study Completion 2014-04-08 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | one year
  The scale measures pain from 0 to 10 and also includes a questionnaire for assessing the activity of daily living.

SECONDARY OUTCOMES:
EuroQol EQ-5D | one year
  The questionnaire measures mobility, ability to care for self, ability to perform usual activities, pain/discomfort, and anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Lewis L Shi, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No